CLINICAL TRIAL: NCT05050578
Title: Clinical Assessment of Two Reusable Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLY935-C022
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Results first posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Refractive Errors
Keywords: Contact lenses
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID018869, then AOHP (Other): Lehfilcon A contact lenses worn in Period 1, followed by senofilcon A contact lenses worn in Period 2, as randomized. Each product will be worn in both eyes during waking hours only for at least 10 hours per day for 30 days. CLEAR CARE will be used for daily contact lens cleaning and disinfection.
  Interventions: Device: Lehfilcon A contact lenses; Device: Senofilcon A contact lenses; Device: CLEAR CARE
- AOHP, then LID018869 (Other): Senofilcon A contact lenses worn in Period 1, followed by lehfilcon A contact lenses worn in Period 2, as randomized. Each product will be worn in both eyes during waking hours only for at least 10 hours per day for 30 days. CLEAR CARE will be used for daily contact lens cleaning and disinfection.
  Interventions: Device: Lehfilcon A contact lenses; Device: Senofilcon A contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: Lehfilcon A contact lenses — Commercially available, silicone hydrogel, spherical contact lenses used as indicated
  Other Names: LID018869
Device: Senofilcon A contact lenses — Commercially available, silicone hydrogel, spherical contact lenses used as indicated
  Other Names: AOHP
Device: CLEAR CARE — Hydrogen peroxide-based contact lens cleaning and disinfecting solution

SUMMARY:
The purpose of this study is to compare the clinical performance of LID018869 soft contact with ACUVUE® OASYS with HYDRACLEAR® PLUS (AOHP) soft contact lenses over 30 days of daily wear.

DETAILED DESCRIPTION:
Subjects will be expected to attend 6 visits. Subjects will be expected to wear their study contact lenses every day for at least 10 hours per day over a 30-day period for each study lens type. The total duration of a subject's participation in the study will be approximately 65 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Current wearer of a commercial spherical weekly/monthly soft contact lenses with at least 3 months of wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day.
* Manifest cylinder less than or equal to 0.75 diopter in each eye.
* Best corrected distance visual acuity better than or equal to 20/25 Snellen in each eye.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Monovision or multifocal lens wearer.
* Habitual senofilcon contact lens wearer (for example, Acuvue Oasys, Acuvue Vita) or commercially available lehfilcon A contact lens wearer (TOTAL30).
* Routinely sleeps in habitual contact lenses.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Vision Care, Study Director — Alcon Research, LLC
Locations (10):
- United States (10):
  - Dr. Elsa Pao, OD, Oakland, California
  - Pacific Rims Optometry, San Francisco, California
  - Sabal Eye Care, Longwood, Florida
  - Vision Health Institute, Orlando, Florida
  - West Bay Eye Associates, Warwick, Rhode Island
  - North Spartanburg Eye Center, Boiling Springs, South Carolina
  - Optometry Group, PLLC, Memphis, Tennessee
  - Advancing Vision Research, LLC, Smyrna, Tennessee
  - Dr Christina R Chang & Associates, OD, PA, Plano, Texas
  - Dawn M. Rakich, OD, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 10 investigative sites located in the United States.
Pre-assignment Details: Of the 166 enrolled, 3 subjects were exited from the study prior to randomization as screen failures, and 1 randomized subject was discontinued prior to exposure to the study lenses. This reporting group includes all subjects exposed to the study lenses, as treated (162).
Units Other Than Participants: eyes
Groups:
- LID018869, Then AOHP: Lehfilcon A contact lenses worn in Period 1, followed by senofilcon A contact lenses worn in Period 2, as randomized. Each product was worn in both eyes during waking hours only for at least 10 hours per day for 30 days. CLEAR CARE was used for daily contact lens cleaning and disinfection.
- AOHP, Then LID018869: Senofilcon A contact lenses worn in Period 1, followed by lehfilcon A contact lenses worn in Period 2, as randomized. Each product was worn in both eyes during waking hours only for at least 10 hours per day for 30 days. CLEAR CARE was used for daily contact lens cleaning and disinfection.
Period: Period 1, 30 Days
Arm/Group | LID018869, Then AOHP | AOHP, Then LID018869
Started | 82; 164 eyes | 80; 160 eyes
Completed | 80; 160 eyes | 79; 158 eyes
Not Completed | 2; 4 eyes | 1; 2 eyes
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2, 30 Days
Arm/Group | LID018869, Then AOHP | AOHP, Then LID018869
Started | 80; 160 eyes | 79; 158 eyes
Completed | 80; 160 eyes | 78; 156 eyes
Not Completed | 0; 0 eyes | 1; 2 eyes
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects exposed to any study lenses.
Groups:
- Total: Total of all reporting groups
Arm/Group | LID018869, Then AOHP | AOHP, Then LID018869 | Total
Number analyzed (Participants) | 82 | 80 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (8.2) | 33.1 (8.5) | 32.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 49 | 94
  Male | 37 | 31 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 70 | 69 | 139
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 56 | 55 | 111
  Black or African American | 5 | 5 | 10
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 18 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 0 | 1
  Multi-racial | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Distance Visual Acuity With Study Lenses at Day 30
Description: Visual acuity (VA) was collected for each eye individually with study lenses in place at a distance of 4 meters using a letter chart. VA was measured in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity.
Time Frame: Day 30, each study lens type
Population: Full Analysis Set: All randomized subjects who were exposed to any study lenses evaluated in this clinical study with data at Day 30.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- LID018869: Lehfilcon A contact lenses worn in Period 1 or Period 2, as randomized, in both eyes during waking hours only for at least 10 hours per day for 30 days. CLEAR CARE was used for daily contact lens cleaning and disinfection.
- AOHP: Senofilcon A contact lenses worn in Period 1 or Period 2, as randomized, in both eyes during waking hours only for at least 10 hours per day for 30 days. CLEAR CARE was used for daily contact lens cleaning and disinfection.
Arm/Group | LID018869 | AOHP
Number analyzed (Participants) | 156 | 158
Number analyzed (eyes) | 312 | 316
logMAR | -0.07 (0.006) | -0.07 (0.006)
Statistical Analysis 1: Comparison: LID018869 vs AOHP; Test type: Non-Inferiority — Noninferiority in distance VA was declared if upper confidence limit was less than 0.05; Since a noninferiority hypothesis is being tested, a p-value is not applicable. Confidence limit is being reported and compared to the noninferiority margin; Least Squares Mean Difference = -0.00, 95% CI 1-sided [upper limit 0.00], Standard Error of Mean 0.003 — LSM results based on mixed effects repeated measures model with both fixed (lens, visit, lens by visit interaction, period, sequence) and random (subject) effects. Difference = LID18869 minus AOHG. Sign is retained with the rounded value

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent to study exit, approximately 65 days.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses, as treated.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses.
- LID018869 Ocular; AOHP Ocular: Events reported in this group occurred while exposed to the lehfilcon A contact lenses.
- LID018869 Non-Ocular; AOHP Non-Ocular: Events reported in this group occurred while exposed to the senofilcon A contact lenses.
Arm/Group | Pretreatment | LID018869 Ocular | LID018869 Non-Ocular | AOHP Ocular | AOHP Non-Ocular
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/322 | 0/161 | 0/320 | 0/160
Serious Adverse Events (participants affected / at risk) | 0/162 | 0/322 | 0/161 | 0/320 | 0/160
Other Adverse Events (participants affected / at risk) | 0/162 | 0/322 | 0/161 | 0/320 | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study,

DOCUMENTS (2):
  • Study Protocol (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT05050578/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT05050578/SAP_001.pdf